CLINICAL TRIAL: NCT00369889
Title: A Phase II Study of Erlotinib Plus Bevacizumab in the Treatment of Advanced Thymoma and Thymic Carcinoma
Brief Title: A Study to Test the Safety and Efficacy of Erlotinib Plus Bevacizumab to Treat Advanced Thymoma and Thymic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUCRO-0148 / 0606-20; AVF3891s (Other: Genentech); IUCRO-0148 (Other: IU Simon Cancer Center)
Record Dates: First submitted 2006-08-28; First posted 2006-08-30 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Thymic Cancer; Thymoma
Keywords: Thymoma; Thymic Cancer
MeSH Terms: conditions — Thymus Neoplasms; Thymoma | interventions — Bevacizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: bevacizumab — iv every 21 days
  Other Names: avastin
Drug: Erlotinib — oral daily
  Other Names: Tarceva

SUMMARY:
The purpose of this study is to determine the rate of response with the combination of erlotinib and bevacizumab in previously treated patients with thymoma or thymic carcinoma, and to determine potential molecular markers that may predict response to therapy in patients with thymoma or thymic carcinoma.

DETAILED DESCRIPTION:
We believe that both the EGFR pathway, as well as tumor angiogenesis play an important role in the pathogenesis of thymic neoplasms. Our previous experience with the EGFR inhibitor gefitinib showed a promising, though limited activity in this disease. We hypothesize that combining the novel EGFR inhibitor erlotinib with bevacizumab will have a synergistic effect on this tumor. We have selected the 15mg/kg q21 days of bevacizumab based on the data published by Johnson DH et al, in which 99 patients were randomly assigned to bevacizumab 7.5 (n = 32) or 15 mg/kg (n = 35) plus carboplatin (area under the curve = 6) and paclitaxel (200 mg/m2) every 3 weeks or carboplatin and paclitaxel alone (n = 32). The highest response noted in the high-dose group (31.5%) and 28.1% in the lower dose bevacizumab arm. There was also a trend to improved TTP and OS in the high dose arm, although the study lacked sufficient power to make any definitive conclusions regarding a possible relationship between dose and treatment effect. (105) The safety and efficacy of this dose and schedule was confirmed by E4599 (43). Herbst et al have confirmed the safety of the combination of erlotinib 150 mg/day orally plus bevacizumab 15 mg/kg in a published phase I/II trial (74)

This regimen has the potential to provide a new, effective therapy for this malignancy, as well as teaching us important lessons about the biology of the disease. To this end, we would also measure surrogate markers of angiogenesis, such as tumor VEGF expression, serum VCAM-1 and bFGF, as well as urine VEGF. We would also determine tumor expression of phosphorylated EGFR, and analyze the effect of known variant polymorphisms in the VEGF gene on outcomes. We will test tumor samples for expression of EGFR by IHC and FISH to correlate to response.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive, recurrent or metastatic thymoma or thymic carcinoma not amenable to potentially curative therapy by surgery in the opinion of the investigator. Original biopsy of tumor is sufficient for diagnoses unless otherwise clinically indicated.
* Patients must have measurable disease per RECIST. Note: Any scans or x-rays used to document measurable disease must be obtained within 28 days prior to registration.
* Patients must have had prior chemotherapy (no limit for prior regimens) for metastatic disease.
* Patients must not have had any form of systemic anticancer therapy within 21 days prior to being registered for protocol therapy.
* Patients receiving radiation therapy must have completed their radiation at least 21 days prior to being registered for protocol therapy, and toxicities due to radiation must have recovered to ≤ grade 1 or baseline prior to registration. Previously radiated area(s) must not be the only site of disease.
* Be at least 18 years of age at the time of consent.
* Patient's must have laboratory data as specified below within 14 days of registration to study:

  1. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times upper limit of normal (ULN) (unless liver metastases are present, in which case AST/ALT ≤ 5 times upper limit of normal will be acceptable).
  2. Total bilirubin ≤ 1.5 mg/dl.
  3. White blood cell (WBC) count > 3000/mm3
  4. Absolute neutrophil count (ANC) ≥ 1500/mm3
  5. Platelets ≥ 100,000/mm3
  6. International normalized ration (INR) of prothrombin time ≤ 1.2, and aPTT no more than 5 seconds longer than the ULN
  7. Urine protein:creatinine ratio 1.0 at screening.
* Patients must not have prior history of malignancy in the past 5 years with the exception of basal cell and squamous cell carcinoma of the skin. Other cancers with low potential for metastasis, such as in situ cancers (e.g., Grade 1, TA TCC (low grade superficial bladder cancer), colonic polyp with focus of adenocarcinoma) can also be enrolled after approval from the study chair.
* No prior use of an EGFR inhibitor or anti-angiogenic agent.
* No use of an investigational agent within 30 days prior to registration for study protocol.
* Must not have any contraindications to the use of erlotinib or bevacizumab as per the package labeling for either product.
* No uncontrolled hypertension ( e.g. > 150/100 mmHg pretreatment)
* No history of unstable angina.
* No history of New York Heart Association (NYHA) Grade II or greater congestive heart failure
* No history of myocardial infarction or angina pectoris/ anginal equivalent in the last 6 months (the patient may be on anti-anginal medications if the symptoms have been entirely controlled for greater than 6 months )within 6 months prior to registration for protocol therapy.
* No history of stroke within 6 months prior to registration for protocol therapy.
* No clinically significant peripheral vascular disease.
* No evidence of bleeding diathesis or coagulopathy.(Low dose anticoagulant therapy to maintain patency of a vascular access device is allowed).
* Patients must not have been using aspirin (>325 mg/day) or another nonsteroidal anti-inflammatory medications known to inhibit platelet function daily within 10 days prior to registration..
* Patients may not be taking the following drugs known to inhibit platelet function: dipyridamole (Persantine), ticlopidine (Ticlid), clopidogrel (Plavix) and cilostazol (Pletal).
* No known evidence of central nervous system involvement or brain metastases. If symptomatic must be confirmed by Head CT or Brain MRI within 6 weeks prior to being registered for protocol therapy.
* No major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to registration for protocol therapy.
* No anticipation of need for major surgical procedure during the course of the study.
* No minor surgical procedures such as fine needle aspirations or core biopsies within 7 days prior to registration for protocol therapy.
* No history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to registration for protocol therapy.
* No serious, non-healing wound, ulcer, or bone fracture.
* No history of hemoptysis.
* No history of deep vein thrombosis or pulmonary embolism.
* No active infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-08; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To determine the objective response rate of the combination of erlotinib and bevacizumab in using RECIST. | completion of study

SECONDARY OUTCOMES:
To determine the time to progression of patients previously treated with thymoma and thymic carcinoma treated with the combination of erlotinib and bevacizumab. | completion of study
To determine the toxicity of the combination of erlotinib and bevacizumab in this patient population. | completion of study
To correlate expression of VEGF in primary tumor sample, circulating VCAM-1 and bFGF, urine VEGF levels pre-therapy with response to therapy. | completion of study
To assess for the effect of known (functionally accepted) variant polymorphisms in the VEGF gene on outcomes. | completion of study
To determine expression of phosphorylated EGFR receptor in tumor specimen | completion of study
To correlate expression of EGFR by IHC and FISH with response to therapy. | completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J Loehrer, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Cancer Center, Indianapolis, Indiana, United States